CLINICAL TRIAL: NCT03615625
Title: Effect of a Power Training Session on Ambulatory Blood Pressure in Older Adults With Hypertension: a Randomized Crossover Trial
Brief Title: Post-exercise Hypotension After a Power Training Session in Older Adults With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 85210618.1.0000.5327
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Exercise; Aging; Ambulatory Blood Pressure Monitoring; Power Exercise
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial with crossover design was performed in order to evaluate the effect of a power training session on office and 24h ambulatory blood pressure in older adults with hypertension.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization list was generated by an epidemiologist using a computer software. This epidemiologist did not participate in the recruitment or assignment to the experimental sessions. Participants and the research team were blinded to the randomization list until the moment of assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control session (No Intervention): Control session without any exercise. The participants remained in seated rest throughout 40 min
- Power Training Session (Experimental): The power training session lasted 40 min, in which the participants performed a resistance exercise session using high velocity contractions during the exercises characterizing a power training session
  Interventions: Behavioral: Power Training Session

INTERVENTIONS:
Behavioral: Power Training Session — 3 sets of 8-10 repetitions of 5 exercises performed in the following order: leg press, bench press, knee extension, upright row, and knee flexion, using an intensity corresponding to 50 % of 1-RM and two-minute intervals between sets and exercises. The concentric phase of exercises during each repetition was performed "as fast as possible" while the eccentric phase lasted 1-2 seconds.
  Arms: Power Training Session

SUMMARY:
The main purpose of the present study was to evaluate the effect of a power training session on office and 24h ambulatory blood pressure in older adults with hypertension. As secondary outcomes, the investigators compared post-exercise hypotension, BP variability, and endothelial function between older men and women with hypertension.

The working hypothesis was that a single bout of power exercise would decrease both office and 24 h BP in comparison to a non-exercising control session and men and women would respond differently after a power training session.

DETAILED DESCRIPTION:
Participants randomly performed two experimental sessions: power exercise training (PT) and non-exercising control at seated rest (Con). They maintained their current antihypertensive medications throughout the trial. Each session was composed of 20 min of rest in the supine position, 40 min of PT or Con protocols, and 60 min of rest in supine position after protocols. The PT was composed of 3 sets of 8-10 repetitions of 5 exercises performed in the following order: leg press, bench press, knee extension, upright row, and knee flexion, using an intensity corresponding to 50 % of 1-RM and two-minute intervals between sets and exercises. The concentric phase of exercises during each repetition was performed "as fast as possible" while the eccentric phase lasted 1-2 seconds. During the Con, the participants remained seated rest on the same exercise machines, but without any exercise. Standardized office BP was performed before and during the first hour (in intervals of 15 min) after exercise and control sessions. Together with the office BP evaluation in the pre and post sessions, the endothelium-dependent brachial vascular function was evaluated using Flow-mediated dilation. Afterwards, participants underwent 24h ambulatory BP monitoring..

ELIGIBILITY:
Inclusion Criteria:

* Office blood pressure between 130-179 and 80-110 mmHg for systolic and diastolic blood pressure, respectively;
* Non-engaged in structured programs of exercise for the last 3 months since the beginning of this study;
* Able to perform the proposed exercises.

Exclusion Criteria:

* Underlying cardiovascular disease previously diagnosticated by a doctor, occurred in the last 24 months, such as: acute myocardial infarction, angina, stroke or heart failure;
* Diseases that reduce life expectancy;
* Smokers and ex-smokers for less than six months;
* BMI > 39.9 kg/m²
* diabetic proliferative retinopathy.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring | 24 hours after control and power training exercise session
  Mean 24-h, day-time, night-time of blood pressure in mmHg will be assessed after each experimental session (power training session and control session)

SECONDARY OUTCOMES:
Office Systolic Blood Pressure | 60 minutes after control and power training exercise session
  Systolic blood pressure in mmHg will be measured using automatic oscillometric before and after each experimental session throughout one hour
Office Diastolic Blood Pressure | 60 minutes after control and power training exercise session
  Diastolic blood pressure in mmHg will be measured using automatic oscillometric before and after each experimental session throughout one hour
Endothelial Function | 60 minutes after control and power training exercise session
  Flow-mediated dilatation (FMD) assessed through high resolution ultrasonography before and after each experimental session throughout one hour
Blood Pressure Variability | 24 hours after control and power training exercise session
  Systolic and diastolic BP values obtained in the 24-hour ambulatory blood pressure monitoring, with valid measures included in a programmed software to calculate the average real variability of these measures.

OTHER OUTCOMES:
Sex Differences in Ambulatory Blood Pressure Monitoring, Office Blood Pressure, Endothelial Function and Blood Pressure Variability | 60 minutes and 24 hours after control and power training exercise session

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ferrari, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Oliveira Carpes L, Domingues LB, Schimitt R, Fuchs SC, Alhalimi T, Tanaka H, Ferrari R. Sex Differences in Post-exercise Hypotension, Ambulatory Blood Pressure Variability, and Endothelial Function After a Power Training Session in Older Adults. Front Physiol. 2021 Jul 16;12:657373. doi: 10.3389/fphys.2021.657373. eCollection 2021. PMID 34335289